CLINICAL TRIAL: NCT03669250
Title: A Placebo-Controlled Study to Evaluate the Effect of a Single Dose of CVN058 on Mismatch Negativity in Subjects With Stable Schizophrenia
Brief Title: CVN058 Effect on Mismatch Negativity in Schizophrenics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevance Alpha, Inc. (Industry)
Responsible Party: Sponsor
Organization: Cerevance (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVN058-103
Record Dates: First submitted 2018-09-04; First posted 2018-09-13 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-07

CONDITIONS: Schizophrenia
Keywords: MMN; EEG; P50; gamma power; P300; auditory gating
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Male and female subjects with schizophrenia, age 18 to 50 years old, inclusive, will be randomized to 1 of 6 treatment sequences to receive 1 of 3 dose regimens in each period; a single oral administration of CVN058, or a matching placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind, placebo controlled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CVN058, low dose (Active Comparator): CVN058 prepared in concentrations of 10mg/mL, and are compounded by the clinical site. Subjects will receive one dose of CVN058 at 15mg or 75mg substitution of 15mg.
  Interventions: Drug: CVN058
- CVN058, high dose (Active Comparator): CVN058 prepared in concentrations of 10mg/mL, and are compounded by the clinical site. Subjects will receive one dose of CVN058 at 150mg.
  Interventions: Drug: CVN058
- Placebo (Placebo Comparator): Matching placebo.
  Interventions: Other: Placebo comparator

INTERVENTIONS:
Drug: CVN058 — CVN058 will be given at two doses, a low does and a high dose
  Other Names: TAK058
  Arms: CVN058, high dose; CVN058, low dose
Other: Placebo comparator — inactive placebo
  Arms: Placebo

SUMMARY:
This is a phase 1, double-blind, placebo-controlled, 3 period cross-over study to evaluate CVN058 target engagement by measuring auditory evoked potential mismatch negativity (MMN) downstream to 5-hydroxytryptamine receptor 3 (5-HT3) as a pharmacodynamic (PD) marker.

DETAILED DESCRIPTION:
Male and female subjects with schizophrenia, age 18 to 50 years old, inclusive, will be randomized to 1 of 6 treatment sequences (Table 2.a) to receive 1 of 3 dose regimens in each period: a single oral administration of CVN058 (15 mg or 150 mg) or matching placebo. The sequence will determine the order in which a subject will take each of the 3 regimens. Discontinued subjects may be replaced at the discretion of the sponsor so that approximately 20 completed subjects are available for analysis.

The study includes three 1-day treatment periods, with a minimum of 7-day washout, maximum 10 day washout (2 total washouts, after Periods 1 and 2) between periods, and a 7-10 day follow-up call post dosing of the last period. Subjects may be inpatients or outpatients at the discretion of the Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 to 50 years of age, inclusive, at the time of informed consent.
* The subject weighs at least 50 kg and has a body mass index (BMI) between 18 and 40 kg/m2 inclusive at Screening.
* Subject meets schizophrenia criteria as defined by the Diagnostic & Statistical Manual of mental Disorders, 5th Edition (DSM-V).
* Subjects are on a stable dose of antipsychotic medication(s) for at least 2 months prior to - Screening as documented by medical history and assessed by site staff.
* Subject has a Positive and Negative Syndrome Scale (PANSS) total score of <95.

Exclusion Criteria:

* Subject currently receiving treatment with any excluded medication or dietary supplement.
* Subjects who have a history of gastrointestinal disease that would influence the absorption of study drug or have a history of any surgical intervention known to impact absorption (e.g., bariatric surgery or bowel resection).
* Subjects having clinical laboratory evaluations (including clinical chemistry, hematology and complete urinalysis) outside the reference range for the testing laboratory, unless the results are deemed to be not clinically significant (NCS) by the investigator at Screening.
* Subjects with moderate to severe substance use disorder, unstable mood or anxiety disorder.
* Subject has a current diagnosis of a significant psychiatric illness other than schizophrenia per DSM-V and is in an acute phase/episode.
* Subject has clinically meaningful hearing loss.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Kapurch, Study Chair — Cerevance, Inc.
Locations (3):
- United States (3):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - New York State Psychiatric Institute, New York, New York
  - Nathan Kline Institute, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 22 eligible participants with schizophrenia including schizoaffective disorder. Eligible participants were randomized to 6 treatment sequences.
Groups:
- Treatment Sequence ABC: Participants were randomized to receive single oral dose of Placebo in treatment period 1 followed by CVN058 15 milligrams (mg) in treatment period 2 followed by CVN058 150 mg in treatment period 3. Each treatment period was followed by a washout-period of 7 days.
- Treatment Sequence BAC; Treatment Sequence ACB: Participants were randomized to receive single oral dose of CVN058 15 mg in treatment period 1 followed by Placebo in treatment period 2 followed by CVN058 150 mg in treatment period 3. Each treatment period was followed by a washout-period of 7 days.
- Treatment Sequence CAB: Participants were randomized to receive single oral dose of CVN058 150 mg in treatment period 1 followed by Placebo in treatment period 2 followed by CVN058 15 mg in treatment period 3. Each treatment period was followed by a washout-period of 7 days.
- Treatment Sequence BCA: Participants were randomized to receive single oral dose of Placebo in treatment period 1 followed by CVN058 150 mg in treatment period 2 and CVN058 15 mg in treatment period 3. Each treatment period was followed by a washout-period of 7 days.
- Treatment Sequence CBA: Participants were randomized to receive single oral dose of CVN058 150 mg in treatment period 1 followed by Placebo in treatment period 2 and CVN058 15 mg in treatment period 3. Each treatment period was followed by a washout-period of 7 days.
Period: Overall Study
Arm/Group | Treatment Sequence ABC | Treatment Sequence BAC | Treatment Sequence CAB | Treatment Sequence ACB | Treatment Sequence BCA | Treatment Sequence CBA
Started | 3 | 3 | 4 | 4 | 4 | 4
Completed | 3 | 2 | 4 | 3 | 3 | 4
Not Completed | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence ABC | Treatment Sequence BAC | Treatment Sequence CAB | Treatment Sequence ACB | Treatment Sequence BCA | Treatment Sequence CBA | Total
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 4 | 4 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.0 (4.00) | 32.0 (8.54) | 35.0 (6.06) | 39.0 (6.63) | 32.5 (14.15) | 36.3 (8.54) | 35.2 (8.06)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: analysis was divided between elderly (65 and over) and non elderly (18-65)
  Participants
    Female | 1 | 0 | 2 | 2 | 0 | 0 | 5
    Male | 2 | 3 | 2 | 2 | 4 | 4 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 1 | 1 | 1 | 9
  Not Hispanic or Latino | 1 | 1 | 2 | 3 | 3 | 3 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 0 | 2 | 1 | 1 | 1 | 0 | 5
  Black/African American | 1 | 0 | 3 | 3 | 1 | 1 | 9
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Reported | 2 | 0 | 0 | 0 | 1 | 0 | 3
  Other | 0 | 1 | 0 | 0 | 1 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean Amplitude of Duration of Auditory Mismatch Negativity (MMN) by Dose Level
Description: MMN is a pre-attentive auditory component elicited by deviant stimuli in an auditory oddball task. Participants were repeatedly exposed to auditory tones and a small proportion of those tones (the "deviant" stimuli) differ from the others (the "standard" stimuli) in their frequency or duration. Typically, the tones are presented, and the evoked potentials are recorded while participants are engaged on a different task, such as reading. Normally, the occurrence of a deviant stimulus increases the amplitude of the negative component in the evoked potential occurring at around 200 msec. MMN is the difference in amplitude between deviant and standard stimuli responses and considered to represent an aspect of pre-attentive novelty detection.
Time Frame: 1.5 hours post-dose on Day 1
Population: Pharmacodynamic Population consisted of all participants who received study drug and had measurements in both the placebo-dosed period and at least one (1) CVN058-dosed period for at least one (1) electroencephalography (EEG)/evoked response endpoint. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: microvolts
Groups:
- Placebo: Participants were randomized to receive Placebo in each treatment period.
- 15mg CVN058: Participants were randomized to receive CVN058 15 mg in each treatment period
- 75mg CVN058: Participants were randomized to receive CVN058 75 mg in each treatment period.
- 150 mg CVN058: Participants were randomized to receive CVN058 150 mg in each treatment period.
Arm/Group | Placebo | 15mg CVN058 | 75mg CVN058 | 150 mg CVN058
Number analyzed (Participants) | 19 | 13 | 6 | 19
microvolts | -0.551 (0.7303) | -0.749 (0.7260) | -0.386 (0.5682) | -1.084 (0.7632)

2. Secondary Outcome: Number of Participants Reporting Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, associated with liver injury and impaired liver function or any other situations as per medical or scientific judgement. TEAEs are defined as any event with onset during or after the first dose of study treatment (active or placebo)
Time Frame: Screening through 30 days post-dose, up to 58 days
Population: Safety Population consisted of all participants who were randomized and received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 15mg CVN058 | 75mg CVN058 | 150 mg CVN058
Number analyzed (Participants) | 20 | 13 | 8 | 19
Participants
  Any TEAE | 1 | 1 | 1 | 4
  Any SAE | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 58 days from screen through study duration
Description: TEAEs and SAEs has been presented for Safety Population. Safety Population consisted of all participants who were randomized and received study drug.
Arm/Group | Placebo | 15mg CVN058 | 75mg CVN058 | 150 mg CVN058
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/13 | 0/8 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/13 | 0/8 | 0/19
Other Adverse Events (participants affected / at risk) | 1/20 | 1/13 | 1/8 | 4/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | 15mg CVN058 (N=13) | 75mg CVN058 (N=8) | 150 mg CVN058 (N=19)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood glucose abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood sodium abnormal (Investigations) | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/50/NCT03669250/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT03669250/SAP_001.pdf